CLINICAL TRIAL: NCT06535022
Title: Impact of Cyclic, Daytime Enteral Nutrition and Ketogenic Nighttime Fasting on the Incidence of Postoperative Delirium in Critically Ill Patients
Brief Title: DeliKet (Substudy of KetoNiFast Study ID 22-1398_1)
Acronym: DeliKet
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Sandra Emily Stoll, MD, Ass. Professor, University Hospital of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-1398_2
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Delirium; Ketogenic Dieting; Nutrition, Healthy
Keywords: ketogenic diet; cyclic nutrition; postoperative delirium
MeSH Terms: conditions — Delirium; Emergence Delirium

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, monocentric, interventional study
Masking Description: sealed, opaque envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group: Cyclic enteral nutrition with ketogenic nighttime fasting (Experimental): Interventional group: Cyclic enteral daytime nutrition (12 hours) with ketogenic nighttime fasting (12 hours) with supplementation of exogenous ketones (ß-hydroxybutyrate) in the Intensive Care Setting.
  Interventions: Dietary Supplement: Cyclic enteral daytime feeding with ketogenic nighttime fasting and exogenous ketone salt supplementation (ß-hydroxybutyrate)
- Control group: Conventional continuous enteral nutrition (No Intervention): Continuous (24 hours) enteral nutrition in the Intensive Care Setting.

INTERVENTIONS:
Dietary Supplement: Cyclic enteral daytime feeding with ketogenic nighttime fasting and exogenous ketone salt supplementation (ß-hydroxybutyrate) — Nighttime fasting and ß-hydroxybutyrate supplementation
  Other Names: cyclic nutrition with nighttime fasting and exogenous ß-hydroxybutyrate supplementation
  Arms: Interventional group: Cyclic enteral nutrition with ketogenic nighttime fasting

SUMMARY:
Postoperative delirium is a common problem of the critically ill patient and associated with an increased mortality. Intermittent fasting and ketogenesis have been shown to be beneficial for maintaining a circadian rhythm and initiating anti-inflammatory repair mechanisms which could potentially be neuroprotective. However, so far there is little data if cyclic enteral feeding with ketogenic nighttime fasting might be beneficial for reducing the rate of postoperative delirium. The study hypothesis is that equicaloric cyclic enteral feeding (12 hrs) during daytime with ketogenic fasting and exogenous ketone supplementation at nighttime compared to continuous standard enteral nutrition (24 hours) decreases the incidence of postoperative delirium in critically ill patients.

DETAILED DESCRIPTION:
Postoperative delirium remains a common postoperative problem in critically ill patients with a prevalence of up to 20% and even up to 50% in the elderly population. But postoperative delirium has a negative impact on mortality as several studies were able to show in the past. Therefore, aiming for a reduction of postoperative delirium has an important impact on patients' outcome. One helpful tool for avoiding postoperative delirium is maintaining a circadian pattern. Enteral feeding may play an important role here. Healthy humans have a circadian feeding pattern with nighttime fasting. There is increasing evidence that a circadian rhythm of feeding (cyclic feeding) could be beneficial for critical ill patients. Cyclic feeding and fasting are assumed to have positive effects on the gut microbiome resulting in optimization of host responses to gastrointestinal pathogens. Another positive effect of cyclic feeding potentially results from activation of a "fasting response", inducing repair pathways such as ketogenesis, mitochondrial biogenesis, anti-inflammatory pathways, antioxidant defenses and autophagy processes. The activation of these repair pathways could diminish cellular stress and promote cellular recovery in critical ill patients. This could have a positive effect on postoperative delirium. A randomized controlled trial by van Dyck et al. could show that fasting-mimicking intervals of 12 hours are sufficient to generate a metabolic fasting response without risking a caloric deficit. This fasting response can be enhanced by additional supplementation of exogenous ketones. The study objective is that equicaloric cyclic enteral feeding (for 12 hours) during daytime with ketogenic fasting (for 12 hours) at nighttime (aiming for a ß-hydroxybutyrate blood concentrations ≥ 0.5mM by exogenous ketone supplementation) compared to continuous (for 24 hours) standard enteral nutrition as per patients' nutritional requirements decreases the incidence of postoperative delirium of critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admission to an ICU
* Start of enteral nutrition

Exclusion Criteria:

* Severe liver insufficiency / liver disease (Child Pugh > B or 7-9 points)
* Post total Pancreatectomy / Insulin-depending diabetes mellitus (IDDM)
* Pregnancy / Lactation
* Hemoglobin-concentration < 80g/l
* Severe metabolic disorder / severe autoimmune disease
* Refractory respiratory or metabolic acidosis
* Disorder of mitochondrial transportation of fatty acids
* Disorder of the oxidation of fatty acids
* Disorder of gluconeogenesis, der ketone body production or ketone body degradation
* Intermittent porphyria
* Severe arrhythmia / cardiomyopathy
* Contraindications against enteral nutrition
* Missing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Confusion Assessment Method (CAM- ICU) | Day 1-14 after randomization or until ICU discharge
  CAM ICU score (lowest score 0, highest score 7)
  • Cognitive function (MoCA- and MMST- Score) day 1, 7, 14 / ICU discharge
• Montreal Cognitive Assessment (MoCA- Score) | Day 1-14 after randomization or until ICU- discharge
  • Cognitive function (MoCA- Score) (lowest Score 0, highest Score 30)
MMSE (Minimental State Examination) | Day 1-14 after randomization or until ICU discharge
  MMSE Score (lowest Score 0, highest Score 30)

SECONDARY OUTCOMES:
Duration of ventilation | From day of randomization until ICU discharge up to 1 month
  Length of invasive and noninvasive ventilation
Length of ICU- and Hospital stay | From day of randomization until hospital discharge up to 6 months
  Length of ICU- and Hospital stay
30-day mortality | From day of randomization up until 30 days
  Mortality at day 30 after ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Bernd W Böttiger, Prof, Study Director — University Hospital Cologne

IPD SHARING:
Plan to Share IPD: No